CLINICAL TRIAL: NCT01296347
Title: A Double-blind, Randomised Placebo-controlled Trial to Determine Whether Low-dose Intravenous Ketamine Peri-operatively Can Prevent Chronic Post-surgical Pain, in Patients Undergoing Thoracotomy or Video Assisted Thoracic Surgery (VATS)
Brief Title: Low Dose Peri-operative IV Ketamine for Chronic Post-surgery Pain Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Gillian Chumbley, Consultant Nurse, Imperial College Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Chumbley1
Record Dates: First submitted 2011-01-31; First posted 2011-02-15 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Chronic Postoperative Pain
Keywords: Ketamine; Thoracotomy; VATS; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (No Intervention): Patients will receive a placebo infusion of 0.9% sodium chloride, which will start 10 minutes prior to the start of the operation and continue for 96 hours.
- ketamine (Experimental): Patients will receive intravenous ketamine, starting 10 minutes prior to surgery and will continue for 96 hours
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intravenous infusion of ketamine starting 10 minutes prior to surgery and running for 96 hours, which will be administered at a rate of 0.1mg/kg/hour. A loading dose of 0.1mg/kg will be administered prior to the start of the infusion
  Other Names: Ketalar
  Arms: ketamine

SUMMARY:
This study will test the null hypothesis that low-dose ketamine given peri-operatively will have no effect on the development of chronic post-surgical pain, in patients undergoing thoracotomy or video assisted thoracic surgery (VATS) procedures

A double-blind, randomised placebo-controlled trial will be used to test the null hypothesis. Potential participants due to undergo either thoracotomy or video assisted thoracic surgery (VATS) will be identified by the collaborating thoracic surgeons in the out-patient department. Patients will be sent information about the study by post, prior to admission for surgery. If they are willing to participate, written consent will be sought on the ward preoperatively, where they will complete baseline measures of pain.

Patients will be randomised to receive an intravenous infusion of placebo (saline) or ketamine running at 0.1mg/kg/hour, starting 10 minutes prior to the surgical incision and continuing for the first three postoperative days (96 hours in total). Prior to starting the infusion a loading dose of ketamine (0.1 mg per kg) will be administered.

DETAILED DESCRIPTION:
This study will test the null hypothesis that low-dose ketamine given peri-operatively will have no effect on the development of chronic post-surgical pain, in patients undergoing thoracotomy or video assisted thoracic surgery (VATS) procedures

A double-blind, randomised placebo-controlled trial will be used to test the null hypothesis. Potential participants due to undergo either thoracotomy or video assisted thoracic surgery (VATS) will be identified by the collaborating thoracic surgeons in the out-patient department. Patients will be sent information about the study by post, prior to admission for surgery. If they are willing to participate, written consent will be sought on the ward preoperatively, where they will complete baseline measures of pain.

Patients will be randomised to receive an intravenous infusion of placebo (saline) or ketamine running at 0.1mg/kg/hour, starting 10 minutes prior to the surgical incision and continuing for the first three postoperative days (96 hours in total). Prior to starting the infusion a loading dose of ketamine (0.1 mg per kg) will be administered. All staff, including the anaesthetist, surgical team, ward nurses and the principal investigator will be blind to the treatment given throughout the study. The key to the randomisation will be revealed at the end of the study.

Patients will be asked to complete a numeric pain score (NPS) and standard pain questionnaires which includes the Brief Pain Inventory [BPI], short form Leeds Assessment of Neuropathic Symptoms and Signs [S-LANSS]) prior to surgery, then at 6 weeks, 3, 6 and 12 months after surgery. The surgical area will also be examined at 6 weeks, 6 and 12 months for signs of neuropathic or nerve pain. Whilst in hospital patients will be asked to score their pain daily, on a numeric pain scale of 0 to 10. Consumption of morphine and side-effects will be recorded.

Patients will receive standard post-operative analgesia.

A sample size calculation based on a previous study, to detect a reduction in pain of 2 points the 10 point numeric pain scale at the 6 week assessment, with α = 5%, 1 - β = 90% and a bilateral hypothesis, would require a sample size of 36 per group, 72 patients in total. This will require a total study population of 144 patients, as both video assisted thoracic surgery (VATS) and thoracotomy patients will be studied.

A two samples t-test will be used to compare the numeric pain scores between the ketamine and placebo groups at each time point. If these data are not normally distributed then the Mann Whitney test will be used. The scores from the Brief Pain Inventory (BPI) and short form Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) will be analysed in the same manner. The Chi Squared test will be used to compare dichotomous data, such as the incidence of side-effects.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years and above) who are undergoing either thoracotomy or video assisted thoracic surgery (VATS).
* Participants must be able to understand English.

Exclusion Criteria:

* Patient refusal
* History of previous chronic thoracic pain
* Neuropathic pain (whatever the site), existing at time of recruitment
* Pre-operative analgesic treatments which include the following medications: strong opioids (step 3 analgesics), tricyclic antidepressants, venlafaxine, gabapentin, pregabalin, duloxetine, clonazepam or carbamazepine.
* Allergy to bupivacaine, morphine, paracetamol, tramadol, dihydrocodeine or ketamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gillian M Chumbley, BSc, PhD, Principal Investigator — Imperial Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chumbley GM, Thompson L, Swatman JE, Urch C. Ketamine infusion for 96 hr after thoracotomy: Effects on acute and persistent pain. Eur J Pain. 2019 May;23(5):985-993. doi: 10.1002/ejp.1366. Epub 2019 Feb 4. PMID 30719817

RESULTS

PARTICIPANT FLOW:
Period: Allocation
Arm/Group | Saline | Ketamine
Started | 38 | 39
Completed | 35 | 35
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — not received infusion | 1 | 0
Period: 6 Week Follow up
Arm/Group | Saline | Ketamine
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: 3 Month Follow up
Arm/Group | Saline | Ketamine
Started | 35 | 34
Completed | 34 | 33
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: 6 Month Follow up
Arm/Group | Saline | Ketamine
Started | 34 | 33
Completed | 32 | 31
Not Completed | 2 | 2
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: 12 Month Follow up
Arm/Group | Saline | Ketamine
Started | 32 | 31
Completed | 28 | 28
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Ketamine | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Full Range); unit: years] | 68 [48 to 87] | 61 [26 to 77] | 64.5 [26 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 12 | 20 | 32
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on Moving at 6 Weeks
Description: Measures in pain include:
  Numeric pain score of 0 to 10. Zero denotes 'no pain'; 10 denotes 'pain as bad as you can imagine'
Time Frame: 6 weeks after surgery
Population: Ketamine group one participant did not have data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Saline: Patients received a placebo infusion of 0.9% sodium chloride, which started 10 minutes prior to the start of the operation and continued for 96 hours.
- Ketamine: Patients received intravenous ketamine, starting 10 minutes prior to surgery and continued for 96 hours
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 35 | 34
units on a scale | 0 [0 to 0] | 1.5 [0 to 4]
Statistical Analysis 1: Comparison: Saline vs Ketamine; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Analgesic Consumption (Opioid)
Description: Analgesia consumption will be measured post-operatively and at 6 weeks
Time Frame: 6 weeks, 3 month, 6 month
Population: Participant who experienced pain.
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- Saline: Patients received a placebo infusion of 0.9% sodium chloride, which started 10 minutes prior to the start of the operation and continue for 96 hours.
- Ketamine: Patients received intravenous ketamine, started 10 minutes prior to surgery and continued for 96 hours
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 18 | 18
mg
  6 weeks | 9 [0 to 26] | 0 [0 to 21]
  3 months | 21 [9 to 47] | 17 [17 to 17]
  6 months | 34 [34 to 34] | 9 [9 to 9]
Statistical Analysis 1: Comparison: Saline vs Ketamine; 6 weeks; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Saline vs Ketamine; 3 month; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Saline vs Ketamine; 6 months; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Sensory Testing
Description: Hypoaesthesia: light touch of the blunt end of a paintbrush was felt less precisely, than in healthy tissue.
  Hyperalgesia: the pain induced by a sterile neurotip, applied perpendicular to the skin is felt abnormally strongly, in comparison to the contralateral side.
  Static allodynia: the application of a Von Frey hair number 14. (8g) was unpleasant, in comparison to the contralateral side.
  Dynamic allodynia: three successive gentle strokes of an 8 mm-wide paintbrush over a 40 mm distance, is unpleasant, in comparison to the contralateral side.
Time Frame: 6 weeks, 6 months, 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Side-effects, Nausea
Description: The presence of nausea recorded at the above time points
Time Frame: 108 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 35 | 35
Participants | 14 | 17
Statistical Analysis 1: Comparison: Saline vs Ketamine; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Incidence of Side Effect, Vomiting
Description: The presence of vomiting recorded at the above time points
Time Frame: 108 hours
Measure: Count of Participants; unit: Participants
Groups:
- Saline: Patients received a placebo infusion of 0.9% sodium chloride, which started 10 minutes prior to the started of the operation and continue for 96 hours.
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 35 | 35
Participants | 8 | 8
Statistical Analysis 1: Comparison: Saline vs Ketamine; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Incidence of Side Effect, Lightheaded
Description: The presence of lightheaded recorded at the above time points
Time Frame: 108 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 35 | 35
Participants | 5 | 14
Statistical Analysis 1: Comparison: Saline vs Ketamine; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Incidence of Side Effect, Vivid Dreams
Description: The presence of vivid dreams recorded at the above time points
Time Frame: 108 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Ketamine
Number analyzed (Participants) | 35 | 35
Participants | 2 | 13
Statistical Analysis 1: Comparison: Saline vs Ketamine; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: For 108 hours the ketamine or placebo infusion was running and whilst the patient remained in hospital after surgery
Arm/Group | Saline | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 8/38 | 9/39
Other Adverse Events (participants affected / at risk) | 34/38 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=38) | Ketamine (N=39)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient developed respiratory distress after thoracotomy, re-intubated and ventilated
Lung hypoinflation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Lung collapse following thoracotomy for cancer, unable to oxygenate. Death due to respiratory failure.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Injury post thoracotomy intubation, causing hoarse voice
Hallucination, visual (Eye disorders) | 2 (2) | 2 (2) — Hallucinations experienced post-operatively, mostly thought to be due to opioids
Confusion postoperative (Psychiatric disorders) | 0 (0) | 0 (0)
Agitation postoperative (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient developed renal failure 13 days after starting trial. Renal biopsy showed undetected myeloma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=38) | Ketamine (N=39)
Dizziness (Nervous system disorders) | 5 (8) | 14 (21) — Patients who felt lightheaded after surgery
Vivid dreams (Nervous system disorders) | 2 (2) | 13 (13) — Vivid dreams experienced after surgery
Nausea (Gastrointestinal disorders) | 14 (14) | 17 (17)
Vomiting (Gastrointestinal disorders) | 8 (8) | 8 (8) — Post-operative vomiting
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No